CLINICAL TRIAL: NCT05558995
Title: Effects and Mechanistic Aspects of Ketogenic Diet in Individuals With Major Depressive Disorder: A Pilot Study
Brief Title: Ketogenic Diet Therapy Major Depressive Disorder
Acronym: KETOMDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Elisa M Brietzke, MD,PhD,Professor, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KETOOPEN
Record Dates: First submitted 2021-11-02; First posted 2022-09-29 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
Keywords: Ketogenic Diet; Major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDD patient (Experimental): Male and female participants (N=10) with ages between 18 and 50 have a confirmed diagnosis of major depressive episode, are experiencing a current episode (following DSM-5 criteria),
  Interventions: Other: ketogenic diet

INTERVENTIONS:
Other: ketogenic diet — All the subjects will be instructed by a nutrition professional to have at least 3 meals per day consisting of 20 g to 30 g of carbohydrate in the form of green vegetables and salad, and 80 g to 100 g of protein in the form of meat, fish, fowl, eggs, shellfish and cheese for 12 weeks. Polyunsaturated and monounsaturated fats will also be included in the diet. Micronutrients (vitamins and minerals) will be given to each subject in the form of one capsule per day. The adherence to diet will be confirmed weekly through a food log and urinary ketones assessment using dipstick to ensure that all individuals remain in a ketotic state.

SUMMARY:
This research program will examine the feasibility as assessed through rates of adherence, tolerability, and safety of the ketogenic diet for individuals with Major Depressive Disorder (MDD) who are not achieving symptomatic remission with first line antidepressants such as the Serotonin Selective Inhibitors (SSRIs). Driven by robust data on the benefits of ketogenic diet in epilepsy and by preliminary data in animal models demonstrating its effects on depressive behaviors, there is a hypothesis that ketogenic diet could be useful to treat residual depressive symptoms. As deficits in reward and pleasure (anhedonia) are the most common residual symptoms in MDD individuals with partial response to SSRIs, the ketogenic diet could be a potential adjuvant in the treatment for depression. In addition, a preliminary assessment of neuroplasticity-related biomarkers in the plasma to determine possible biological substrates for the mechanism of action of ketogenic diet in the brain will be conducted.

DETAILED DESCRIPTION:
This is a 12-week, open-label study of the feasibility, safety, and tolerability of adjunctive ketogenic diet for the treatment of individuals with Major Depressive Disorder (MDD). The study will consist of a 2-weeks ketogenic diet induction phase, followed by a 10-week maintenance phase until study endpoint (week-12). For this feasibility study, 15 participants that successfully meet the requirements for inclusion in the study will be enrolled. With an expected patient dropout rate of approximately 15% at 12-weeks, this sample size will be effective in reliably estimating patient adherence and tolerability to the ketogenic diet, and patient recruitment and dropout rates. The results of this feasibility study will facilitate the calculation of an appropriate sample size for a subsequent randomized controlled trial. Research individuals will be recruited from the Mood Disorders Outpatient Unit at Providence Care Hospital and the W.J. Henderson Centre for Patient-Oriented Research at Kingston General Hospital (KGH) both located in Kingston, ON, Canada. Male and female participants with ages between 18 and 50 who have had a confirmed diagnosis of a major depressive episode and currently meeting all inclusion and exclusion criteria, and which are able to provide written informed consent will be eligible for inclusion in the study. A virtual appointment will be arranged for participants interested in participation with research staff members and a registered dietitian also will interview the individual to ensure that participants fully understand the study. Details on the ketogenic diet, the foods involved, and other dietary questions, will be answered by a registered dietician. If complete eligibility is confirmed, patients will be given 48 hours to decide on participation. If willing to participate in the study, written informed consent will be obtained. The study consists in weekly visits involving psychiatric assessments, general medical assessments, and dietetic assessments. The first two will be conducted by trained psychiatrist and the third one by a registered dietician. In every visit the psychiatrists will conduct assessments of severity of depressive symptoms and anhedonia and treatment-emergent side effects. The computer based task Effort Expenditure for Rewards Task (EEfRT) will be used to evaluate reward motivation at the baseline and at the endpoint. Weight, height, Body Mass Index, waist circumference, and hip circumference will be evaluated in all visits. The individuals will be asked to fill a food diary that will be checked at each weekly consultation. The quantities of food will be recorded by each patient. The exact macronutrient consumption will be analyzed and recorded for each patient by the registered dietician. The dietician will analyze all foods and drinks consumed by participants to ensure each individual is abiding to the medically supervised ketogenic diet. Urine will be collected in each visit for assessment of ketonuria, a parameter of adherence to the intervention. A blood sample will be collected at the baseline and endpoint consultations for biological analysis of neuroplasticity-related biomarkers in plasma. The results of this study will demonstrate whether consumption of the medically supervised ketogenic diet for 12 consecutive weeks by individuals with MDD is a feasible and tolerable intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for single episode or recurrent MDD, without psychotic features, according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), and confirmed by the Mini International Neuropsychiatric Interview (MINI).

  -- Moderate or severe depressive syndrome, as defined by a Montgomery-Asberg Depression Rating Scale (MADRS) total score greater than or equal to (>=) 20 at baseline.
* Treatment with SSRIs for at least 6 weeks, with no changes in dosing for the past 3 weeks.
* Must be capable of providing informed consent, based on the opinion of the participating physician.
* No vitamin and mineral deficiencies, specifically: vitamin B (B1, B3, B6, B9, and B12), vitamin D, iron, zinc, electrolytes (Na, K), calcium, and magnesium.

Exclusion Criteria:

* Has a current or prior diagnosis of schizophrenia spectrum disorders or bipolar disorder or related disorders, or intellectual disability, according to DSM-5.
* Has current or prior diagnosis of epilepsy
* Has homicidal ideation/intent or is at imminent risk of suicide per the physician's clinical judgment and/or based on the Columbia-Suicide Severity Rating Scale (C-SSRS) corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent)
* Has received electroconvulsive therapy in the past 6 months. - Made use of caloric restriction, intermittent fasting, and carbohydrates restriction in the 4 weeks prior the inclusion.
* Adoption of specific dietetic habits: vegan, gluten-free, lactose-free diets or currently doing fasting for religious purposes.
* Has evidence of alcohol or drug dependence (except for nicotine and caffeine) according to DSM-5 or within 6 months prior to enrolment
* Has participated in or is currently enrolled in any clinical trial or observational study within the current episode.
* Has a medical contra-indication for ketogenic diet (e.g. metabolic disorder, cardiac arrhythmia, pregnancy or breastfeeding).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Participant Adherence | Baseline (week 0), week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12.
  Number of participants that completed the trial/Total number of participants enrolled

SECONDARY OUTCOMES:
Changes in the Effort-based decision making | Baseline (week 0), week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12.
  the Effort-Expenditure for Rewards Task (EEfRT or "effort"), a novel behavioral paradigm as a means of exploring effort-based decision-making in humans. The proportion of hard-task choices indicates a more active reward system.
Changes in the serum levels of the brain-derived neurotrophic factor | Baseline (week 0) and week 12.
  The BDNF levels will be determined in plasma with the enzyme-linked immunosorbent assay (ELISA), as part of the biomarkers assessments. Results are expressed in pg/mL.
Changes in the serum level of TNF-alpha | Baseline (week 0) and week 12.
  The TNF-alpha blood levels will be determined by ultrasensitive ELISA. The results will be expressed in pg/mL.
Changes in the serum level of Interleukin-1(IL-1) | Baseline (week 0) and week 12.
  The IL-1 blood levels will be determined by ultrasensitive ELISA. The results will be expressed in pg/mL.
Changes in the serum level of Interleukin-6 (IL-6) | Baseline (week 0) and week 12.
  The IL-6 blood levels will be determined by ultrasensitive ELISA. The results will be expressed in pg/mL.
Changes in the serum level of Interleukin-6 (IL-10) | Baseline (week 0) and week 12.
  The IL-10 blood levels will be determined by ultrasensitive ELISA. The results will be expressed in pg/mL.
Changes in depressive symptoms severity | Baseline (week 0), week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12.
  Montgomery-Asberg Depression Rating Scale to assess changes in severity of depressive symptoms. The scores of this scale varies from 0-60 with higher scores indicating more severe depressive symptoms.
Changes in anxiety symptoms severity | Baseline (week 0), week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12.
  Generalized Anxiety Disorder-7 to assess severity of anxiety symptoms. The scores in this instrument vary from 0-21 with higher scores indication greater severity of anxiety symptoms.
Changes in functioning | Baseline (week 0), week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12.
  Clinical Global Impression. The score of this scale varies from 1-7, with higher scores indicating poorer functioning
complete blood count (CBC) baseline | Baseline (week 0)
  complete blood count (CBC) as part of safety assessment
complete blood count (CBC) endopoint | Endpoint (week 12)
  complete blood count (CBC) as part of the safety assessment
Sodium blood level baseline | Baseline (week 0)
  Sodium blood level blood expressed in mEq/L as part of the safety assessment
Sodium blood level endpoint | Endpoint (week 12)
  Sodium blood level blood expressed in mEq/L as part of the safety assessment
Potassium blood level baseline | Baseline (week 0)
  Potassium blood level blood expressed in mEq/L as part of the safety assessment
Potassium blood level endpoint | Endpoint (week 12)
  Potassium blood level blood expressed in mEq/L as part of the safety assessment
Vitamin B blood level baseline | Baseline (week 0)
  Vitamin B blood level expressed in pg/mL as part of the safety assessment
Vitamin B blood level endpoint | Endpoint (week 12)
  Vitamin B blood level expressed in pg/mL as part of the safety assessment
Vitamin D blood level baseline | Baseline (week 0)
  Vitamin D blood level expressed in pg/mL as part of the safety assessment
Vitamin D blood level | Endpoint (week 12)
  Vitamin D blood level expressed in pg/mL as part of the safety assessment
Iron serum level baseline | Baseline (week 0)
  Iron serum level expressed in mcg/dL as part of the safety assessment
Iron serum level endpoint | Endpoint (week 12)
  Iron serum level expressed in mcg/dL as part of the safety assessment
Zinc blood level baseline | Baseline (week 0)
  Zinc blood level expressed in mcg/mL as part of the safety assessment
Zinc blood level endpoint | Endpoint (week 12)
  Zinc blood level expressed in mcg/mL as part of the safety assessment
Blood level of aspartate aminotransferase (AST) baseline | Baseline (week 0)
  Blood level of aspartate aminotransferase (AST) expressed in U/L
Blood level of aspartate aminotransferase (AST) endpoint | Endpoint (week 12)
  Blood level of aspartate aminotransferase (AST) expressed in U/L as part of the safety assessment
Blood level of alanine aminotransferase (ALP) baseline | Baseline (week 0)
  Blood level of alanine aminotransferase (ALP) expressed in U/L as part of the safety assessment
Blood level of alanine aminotransferase (ALP) endpoint | Endpoint (week 12)
  Blood level of alanine aminotransferase (ALP) expressed in U/L as part of the safety assessment
Blood level of albumin baseline | Baseline (week 0)
  Blood level of albumin (ALB) expressed in g/dL as part of the safety assessment
Blood level of albumin endpoint | Endpoint (week 12)
  Blood level of albumin (ALB) expressed in g/dL as part of the safety assessment
Blood prothrombin time (PT) baseline | Baseline (week 0)
  Prothrombin time (PT) expressed in prothrombin time/international normalized ratio (INR) as part of the safety assessment
Blood prothrombin time (PT) endpoint | Endpoint (week 12)
  Prothrombin time (PT) expressed in prothrombin time/international normalized ratio (INR) as part of the safety assessment
Total serum bilirubin baseline | Baseline (week 0)
  Total serum bilirubin expressed in mg/dL as part of the safety assessment
Total serum bilirubin endpoint | Endpoint (week 12)
  Total serum bilirubin expressed in mg/dL as part of the safety assessment
Serum blood urea nitrogen (BUN) baseline | Baseline (week 0)
  blood urea nitrogen (BUN) expressed in mmol/L as part of the safety assessment
blood urea nitrogen (BUN) endpoint | Endpoint (week 12)
  blood urea nitrogen (BUN) expressed in mmol/L as part of the safety assessment
Urinalysis (UA) baseline | Baseline (week 0)
  Urinalysis (UA) for ketonuria as part of the safety assessment
Urinalysis (UA) endpoint | Endpoint (week 12)
  Urinalysis (UA) for ketonuria as part of the safety assessment
Blood glycated hemoglobin (HbA1c) in the baseline | Baseline (week 12)
  Blood glycated hemoglobin (HbA1c), expressed in % as port of the safety assessment
Blood glycated hemoglobin (HbA1c) in the endpoint | Endpoint (week 12)
  Blood glycated hemoglobin (HbA1c), expressed in % as part of the safety assessment
Lipid panel baseline | Baseline (week 0)
  lipid panel as part of the safety assessment
Lipid panel endpoint | Endpoint (week 12)
  lipid panel as part of the safety assessment
Pregnancy test (for female participants) | Baseline (week 0)
  Pregnancy test (for female participants)
Pregnancy test (for female participants) | Endpoint (week 12)
  Pregnancy test (for female participants)
Changes in severity of anhedonia | Baseline (week 0), week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12.
  Snaith-Hamilton Pleasure Scale (SHAPS) to assess severity of anhedonia. The scores varies from 0-14. A higher total score indicates higher levels of anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Brietzke, MD,PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University - Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Currently, we do not have the plan of individual participant data (IPD) sharing. Data transfer outside the institute has to be approved by Institutional Review Board at Queen's University.

REFERENCES:
- [Background] Malhi GS, Mann JJ. Depression. Lancet. 2018 Nov 24;392(10161):2299-2312. doi: 10.1016/S0140-6736(18)31948-2. Epub 2018 Nov 2. PMID 30396512
- [Background] Shelton RC, Tomarken AJ. Can recovery from depression be achieved? Psychiatr Serv. 2001 Nov;52(11):1469-78. doi: 10.1176/appi.ps.52.11.1469. PMID 11684742
- [Background] Cooper JA, Arulpragasam AR, Treadway MT. Anhedonia in depression: biological mechanisms and computational models. Curr Opin Behav Sci. 2018 Aug;22:128-135. doi: 10.1016/j.cobeha.2018.01.024. PMID 29503842
- [Background] Ceolin G, Breda V, Koning E, Meyyappan AC, Gomes FA, Moreira JD, Gerchman F, Brietzke E. A Possible Antidepressive Effect of Dietary Interventions: Emergent Findings and Research Challenges. Curr Treat Options Psychiatry. 2022;9(3):151-162. doi: 10.1007/s40501-022-00259-1. Epub 2022 Apr 23. PMID 35496470
- [Background] Grigolon RB, Gerchman F, Schoffel AC, Hawken ER, Gill H, Vazquez GH, Mansur RB, McIntyre RS, Brietzke E. Mental, emotional, and behavioral effects of ketogenic diet for non-epileptic neuropsychiatric conditions. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Aug 30;102:109947. doi: 10.1016/j.pnpbp.2020.109947. Epub 2020 Apr 17. PMID 32305355
- [Background] Brietzke E, Mansur RB, Subramaniapillai M, Balanza-Martinez V, Vinberg M, Gonzalez-Pinto A, Rosenblat JD, Ho R, McIntyre RS. Ketogenic diet as a metabolic therapy for mood disorders: Evidence and developments. Neurosci Biobehav Rev. 2018 Nov;94:11-16. doi: 10.1016/j.neubiorev.2018.07.020. Epub 2018 Jul 31. PMID 30075165
- [Derived] Brietzke E, Fabe J, Bambokian A, Breda V, Chaves C, Shelp J, Terpstra A, Koning E, Groll D, Milev R, McIntyre RS, Mansur RB, Soares CN, Gomes FA. Medically supervised ketogenic diet as an adjunctive treatment for moderate to severe depression: A pilot study. J Affect Disord. 2026 Apr 15;399:121079. doi: 10.1016/j.jad.2025.121079. Epub 2025 Dec 29. PMID 41475571